CLINICAL TRIAL: NCT00355264
Title: Phase 2, Multicenter, Open Label Study of Phenoptin in Subjects With Hyperphenylalaninemia Due to Primary BH4 Deficiency
Brief Title: Safety and Efficacy Study of Phenoptin in Subjects With Hyperphenylalaninemia Due to BH4 Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-007
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Tetrahydrobiopterin Deficiencies; Hyperphenylalaninemia, Non-Phenylketonuric
MeSH Terms: conditions — Phenylketonurias | interventions — phenoptin

STUDY DESIGN:
Intervention Model Description: Outcomes were to be evaluated for all subjects with primary BH4 disease. Outcomes were also evaluated based on the type of BH4 deficiency either due to defects in the genes encoding the enzymes involved in BH4 biosynthesis, GTPcyclohydrolase I (GCH1), 6-pyruvoyl-tetrahydropterin synthase (PTPS), and sepiapterin reductase (SR); or defects in the genes encoding the enzymes involved in BH4 recycling, pterin-4a-carbinolamine dehydratase (PCD) and dihydropteridine reductase (DHPR)

ARMS (1):
- Single Arm on Active Drug (Experimental): 5mg/kg/day orally, dose may be adjusted to between 5-20 mg/kg/day by investigator at week 6 to control blood Phe levels
  Outcomes were also evaluated by the subject's type of BH4 deficiency either defects in the genes encoding the enzymes involved in biosynthesis or defects in the genes encoding the enzymes involved in recycling.
  Interventions: Drug: Phenoptin

INTERVENTIONS:
Drug: Phenoptin — 5mg/kg/day orally, dose may be adjusted to between 5-20 mg/kg/day by investigator at week 6 to control blood Phe levels

SUMMARY:
The purpose of this study is to evaluate the ability of Phenoptin to control blood phenylalanine levels in subjects who have hyperphenylalaninemia due to a primary BH4 deficiency and to evaluate the safety of Phenoptin in this population. Some subjects were receiving non-registered formulations of BH4 at enrollment and this treatment was suspended after Part 1 and within one day the subjects started Phenoptin at approximately the same dose.

DETAILED DESCRIPTION:
Within 4 weeks of completing screening assessments to determine eligibility, subjects will be enrolled in the study. The study will be conducted in two parts.

Part 1: After screening, all subjects will be followed for two weeks without modification of their baseline medical or dietary care.

Part 2: Beginning at Week 2, subjects who were receiving non-registered formulations of BH4 at enrollment will suspend this treatment and within one day will start Phenoptin at approximately the same dose of the non-registered BH4 formulation. Subjects not receiving BH4 at enrollment will begin treatment with Phenoptin at approximately 5 mg/kg/day, given orally, prior to meals.

At the discretion of the Investigator, the Phenoptin dose may be adjusted up or down at the Week 6 visit to control blood Phe levels (<360 µmol/L), or to optimize the clinical effect. The maximum dose allowed will be approximately 20 mg/kg/day. All subjects will receive Phenoptin for a total of 8 weeks. Subjects will be instructed to continue their usual diet without modification. Study visits will occur every other week.

Tyrosine, biopterin and neopterin will be analyzed at the following visits: Week 0 (enrollment), Week 2 (prior to dosing with Phenoptin), Week 8 (after 6 weeks of treatment with Phenoptin) and Week 10 (after 8 weeks of treatment with Phenoptin).During each visit, blood Phe level will be measured (2.5-5 hours after a meal), and safety evaluations will be performed. Safety will be assessed by monitoring adverse events and vital signs, performing physical examinations, assessing signs and symptoms of primary BH4 deficiency (i.e., neurological symptoms such as seizures, changes in muscle tone, weakness, etc.) and clinical laboratory tests (chemistry, hematology and urinalysis).

Extension: Upon completion of 8 weeks of treatment (i.e., at the Week 10 visit), subjects will be offered the option to continue treatment with Phenoptin in an extension of this study. Participation in the study extension will continue until one of the following occurs:

1. the subject withdraws consent and discontinues from the study,
2. the subject is discontinued from the study at the discretion of the investigator,
3. the study drug is available through the appropriate marketing approval, or
4. the study is terminated.

During the extension period, study drug will be dispensed to subjects monthly, and study visits will be required every 3 months. The Phenoptin dose may be adjusted at any visit during the study extension at the discretion of the Investigator. The maximum dose allowed will be approximately 20 mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of blood Phe level > 180 µmol/L on at least one occasion
* Established diagnosis of hyperphenylalaninemia (HPA) due to primary BH4 deficiency with a documented defect in biopterin metabolism with blood or urine tests
* Willing and able to provide written informed consent or, in the case of subjects under the age of 18 years, provide written assent (if required) and written informed consent by a parent or legal guardian
* Negative urine pregnancy test at screening for females of child-bearing potential
* Male and female subjects of childbearing potential (if sexually active and non-sterile) must be using acceptable birth control measures and be willing to continue to use acceptable birth control measures, as determined by the Investigator, and be willing to continue to use acceptable birth control measures while participating in the study
* Willing and able to comply with all study procedures
* Able to take medication orally

Exclusion Criteria:

* Perceived to be unreliable or unavailable for study participation or, if under the age of 18 years, have parents or legal guardians who are perceived to be unreliable or unavailable
* Use of any investigational agent (other than BH4) within 30 days prior to screening, or requirement for any investigational agent or vaccine prior to completion of all scheduled study assessments
* Positive urine pregnancy test at screening (non-sterile females of child bearing potential only), already known to be pregnant or breastfeeding or planning a pregnancy in self or partner during the study
* Female subjects of childbearing potential not using an effective method of birth control, as determined by the PI, or unwilling to continue to use acceptable birth control measures.
* Alanine aminotransferase (ALT) > 2 times the upper limit of normal (i.e., Grade 1 or higher based on World Health Organization Toxicity Criteria) at screening
* Concurrent disease or condition that would interfere with study participation or safety (e.g., seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, insulin-dependent diabetes, or organ transplantation)
* Serious neuropsychiatric illness (e.g., major depression) not currently under medical control
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (e.g., methotrexate)
* Clinical diagnosis of phenylketonuria (PKU) due to phenylalanine hydroxylase deficiency
* Any condition that, in the view of the PI, renders the subject at high risk from treatment compliance and/or completing the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Los Angeles, California
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - New York, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Salt Lake City, Utah
  - Seattle, Washington
  - Madison, Wisconsin
- Düsseldorf, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicenter study, conducted at 8 sites in the United States of America and one site in Germany
Pre-assignment Details: A sample size planned of 10 to 15 subjects considered adequate based on clinical considerations. Actual enrolled and treated are 12 subjects.
Groups:
- Phenoptin: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of Tetrahydrobiopterin (BH4) at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half of the dose was administered orally twice daily, to achieve a full dose per day.
  In Part 3 (concurrent with Extension), subjects had the option of receiving 10 mg/kg/day Phenoptin administered orally twice daily for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects that completed Part 2 were offered the option of participating in Part 3. Among 12 subjects, 2 participated in Part 3 that took place concurrent with the Extension study.
Period: Part 1 (2 Weeks)
Arm/Group | Phenoptin
Started | 12
Completed | 12
Not Completed | 0
Period: Part 2 (8 Weeks)
Arm/Group | Phenoptin
Started | 12
Completed | 12
Not Completed | 0
Period: Part 3 (7 Weeks of Extension)
Arm/Group | Phenoptin
Started | 2
Completed | 2
Not Completed | 0
Period: Extension (Variable Duration)
Arm/Group | Phenoptin
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Groups:
- Phenoptin: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, administered orally twice for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin.
  The mean Phenoptin dose received during the study was 9.1 mg/kg/day with a minimum of 1.9 mg/kg/day and a maximum of 21 mg/kg/day.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 are offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
Arm/Group | Phenoptin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  <18 years of age | 10
  >=18 and <65 years of age | 2
  >=65 years of age | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 10
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  North America | 10
  Europe | 2
Height [Mean (Standard Deviation); unit: cm] | 142.1 (27.6)
Weight [Mean (Standard Deviation); unit: kg] | 45.2 (27.1)
Type of Enzyme Defects [Number; unit: participants] — Subjects were classified into 2 groups (synthesis and recycling groups) based on the response to a medical history query as to the type of enzymatic defect that caused primary BH4 deficiency in each subject. Nine (75.0%) subjects had defects in enzymes involved in BH4 biosynthesis and formed the synthesis group. Three subjects (25.0%) had defects in enzymes involved in recycling BH4 from an oxidized form back to an active reduced state.
  participants
    Synthesis | 9
    Recycling | 3
Blood Phe at Screening Visit [Mean (Standard Deviation); unit: µmol/L] | 164.5 (186.8)

OUTCOME MEASURES:

1. Primary Outcome: Blood Phenylalanine(Phe) Levels Measured at Specified Timepoints
Description: Baseline blood phenylalanine(Phe) value is the latest measurement taken prior to initiation of Phenoptin treatment. The ideal range for blood Phe levels is approximately 120-360 µmol/L.
Time Frame: At Baseline, Week 4 through Extension Week 130
Population: Efficacy analysis population are the subjects received at least 1 dose of Phenoptin and has at least 1 post-treatment measurement of blood Phe.
Measure: Mean (Standard Deviation); unit: μmol/L
Groups:
- All Subjects: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, half a dose administered orally twice daily for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 are offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
- Subgroup: Subjects With Synthesis Enzymatic Defect: Subjects primary BH4 deficiency due to defects in the genes encoding the enzymes involved in BH4 biosynthesis, guanosine triphosphate (GTP) cyclohydrolase I (GCH1), 6-pyruvoyl-tetrahydropterin synthase (PTPS), and sepiapterin reductase (SR).
- Subgroup: Subjects With Recycling Enzyme Defect: Subjects with BH4 deficiency due to defects in the genes encoding the enzymes involved in BH4 recycling, pterin-4a-carbinolamine dehydratase (PCD) and dihydropteridine reductase (DHPR).
Arm/Group | All Subjects | Subgroup: Subjects With Synthesis Enzymatic Defect | Subgroup: Subjects With Recycling Enzyme Defect
Number analyzed (Participants) | 12 | 9 | 3
μmol/L
  Baseline | 132.9 (134.7) | 72.2 (13.4) | 315.0 (180.9)
  Part 2: Week 4 | 104.1 (66.7) | 78.2 (28.4) | 181.7 (96.1)
  Part 2: Week 6 | 120.8 (119.0) | 70.2 (17.2) | 272.7 (175.1)
  Part 2: Week 8 | 112.3 (106.8) | 66.6 (13.6) | 249.3 (156.2)
  Part 2: Week 10 | 143.2 (147.3) | 75.0 (11.5) | 347.7 (187.7)
  Extension: Week 22 | 94.3 (76.5) | 63.8 (8.5) | 185.7 (123.1)
  Extension: Week 34 | 105.0 (95.3) | 71.9 (16.6) | 204.3 (170.8)
  Extension: Week 46 | 144.8 (164.2) | 78.8 (20.4) | 343.0 (261.0)
  Extension: Week 58 | 151.4 (173.1) | 72.4 (17.7) | 388.3 (226.6)
  Extension: Week 70 | 106.7 (93.8) | 72.0 (12.6) | 210.7 (161.6)
  Extension: Week 82 | 153.0 (223.2) | 61.3 (12.1) | 428.0 (349.4)
  Extension: Week 94 | 186.2 (305.8) | 63.8 (10.6) | 553.3 (494.2)
  Extension: Week 106 | 157.2 (159.8) | 69.8 (21.7) | 419.3 (33.0)
  Extension : Week 118 | 124.3 (119.4) | 73.1 (22.8) | 277.7 (171.1)
  Extension: Week 130 | 124.9 (118.2) | 74.6 (14.9) | 276.0 (173.9)

2. Primary Outcome: Percentage of Subjects With Blood Phenylalanine (Last Observation Carried Forward) < 360 μmol/L
Description: Baseline blood phenylalanine(Phe) value is the latest measurement taken prior to initiation of Phenoptin treatment. The objective of this outcome was to compare to Phe levels achieved using previous treatment regimens.
Time Frame: At Baseline, Week 4 through Extension Week 130
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Subjects: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, administered orally twice for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin, either resumed with previously taken BH4 (tetrahydrobiopterin) formulations.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 are offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
Arm/Group | All Subjects
Number analyzed (Participants) | 12
percentage of participants
  Baseline | 83.3 [51.6 to 97.9]
  Part 2: Week 4 | 100 [73.5 to 100]
  Part 2: Week 6 | 91.7 [61.5 to 99.8]
  Part 2: Week 8 | 91.7 [61.5 to 99.8]
  Part 2: Week 10 | 91.7 [61.5 to 99.8]
  Extension: Week 22 | 100 [73.5 to 100]
  Extension: Week 34 | 91.7 [61.5 to 99.8]
  Extension: Week 46 | 83.3 [51.6 to 97.9]
  Extension: Week 58 | 83.3 [51.6 to 97.9]
  Extension: Week 70 | 91.7 [61.5 to 99.8]
  Extension: Week 82 | 83.3 [51.6 to 97.9]
  Extension: Week 94 | 83.3 [51.6 to 97.9]
  Extension: Week 106 | 75 [42.8 to 94.5]
  Extension: Week 118 | 83.3 [51.6 to 97.9]
  Extension: Week 130 | 83.3 [51.6 to 97.9]

3. Secondary Outcome: Subjects Experiencing Adverse Events(AEs)
Description: Intensity was determined by the Investigator. For symptomatic AEs the following definitions were applied.
  Mild = AE did not limit usual activities.
  Moderate = AE resulted in some limitation of usual activities.
  Severe = AE resulted in an inability to carry out usual activities.
  A treatment-emergent Adverse Events (TEAE) is any Adverse Events that newly appeared, increased in frequency or worsened in severity following initiation of study drug administration.
  Serious AE (SAE) resulted in death, was life-threatening, required in patient hospitalization or prolongation of an existing hospitalization, resulted in persistent or significant disability or incapacity, is a congenital anomaly or birth defect; or was an important medical event.
Time Frame: Up to 35 Months
Measure: Number; unit: participants
Groups:
- Phenoptin: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, administered orally twice for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 are offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
Arm/Group | Phenoptin
Number analyzed (Participants) | 12
participants
  Any Adverse Events | 12
  Study Drug-Related Adverse Events | 6
  Any Serious Adverse Events | 2
  Withdrawal from study due to AE | 1
  Withdrawal from Study due to SAE | 0
  TEAE by severity: Mild | 4
  TEAE by severity: Moderate | 6
  TEAE by severity: Severe | 2

4. Other Pre Specified Outcome: AEs Consistent With Signs and/or Symptoms of BH4 Deficiency
Description: Attention was paid to AEs that may be consistent with signs and/or symptoms associated with primary BH4 deficiency to determine if such signs and symptoms arose or increased in severity or frequency during the study. These included prematurity and low birth weight, inability to control body temperature, low muscle tone, decreased spontaneous movements, poor sucking, movement disorders, difficulty swallowing, hypersalivation, seizures or convulsions, behavioral problems, developmental delay, and mental retardation.
Time Frame: Up to 35 months
Population: AEs that are signs and symptoms of BH4 deficiency were reported for 3 subjects: One SAE of mild dyskinesia (required hospitalization) in one subject; events of severe dystonia and moderate Dyskinesia in one subject; and one event of mild vertigo in one subject. All events resolved and were considered unrelated to Phenoptin except mild vertigo.
Measure: Count of Participants; unit: Participants
Groups:
- Phenoptin: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, administered orally twice for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 were offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
Arm/Group | Phenoptin
Number analyzed (Participants) | 12
Participants
  Subjects with Any Signs and/or Symptoms of BH4 Def | 3
  Dystonia | 1
  Dyskinesia | 2
  Vertigo | 1

ADVERSE EVENTS:
Time Frame: Up to 35 months (from enrollment to Study Completion.)
Groups:
- Phenoptin: In Part 1, subjects continued their usual treatment regimen.
  In Part 2, subjects on non-registered formulations of BH4 at enrollment began Phenoptin treatment at approximately the same daily dose; subjects not receiving BH4 at enrollment began treatment at 5mg/kg/day Phenoptin. Half a dose was administered orally twice daily, to achieve a full dose/day.
  In Part 3, subjects receives 10 mg/kg/day Phenoptin, administered orally twice for three weeks, followed by 20 mg/kg/day once daily for remaining 4 weeks.
  In extension phase, subjects were offered the option to continue treatment with Phenoptin, either resumed with previously taken BH4 (tetrahydrobiopterin) formulations.
  All 12 subjects participated in Part 1, Part 2 and Extension Phase. Subjects completed Part 2 are offered the option of participating in Part 3, Subjects who agreed to participate proceeded to Part 3. Among 12 subjects, 2 participated in Part 3.
Arm/Group | Phenoptin
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenoptin (N=12)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Medical Device Change (Surgical and medical procedures) | 1 (1)
Dyskinesia (Nervous system disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phenoptin (N=12)
Neutropenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 2
Irritability (General disorders) | 1
Pyrexia (General disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 5
Otitis media (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin candida (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral skin infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood calcium increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Metabolic function test abnormal (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Urine ketone body present (Investigations) | 1
Urine leukocyte esterase positive (Investigations) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Skin inflammation (Skin and subcutaneous tissue disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Dyskinesia (Nervous system disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Medical device change (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
Due to the small sample size in this study, a single patient AE exceeded the 5% maximum AE reporting threshold. Many of these manifestations are due to primary BH4 deficiency disease and the associated inadequate neurotransmitters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No